CLINICAL TRIAL: NCT01173614
Title: Project Gullstrand - European Project for the Determination of Average Biometric Values of Human Eyes
Acronym: Gullstrand
Status: Completed | Type: Observational
Sponsor: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: ECR-CCRS-2010-01
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Normal Subjects, Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal subjects: Subjects with two normal eyes.

SUMMARY:
The purpose of this study is to determine the average values of human ocular biometry and to correlate these values with visual function.

ELIGIBILITY:
Inclusion Criteria:

* Two normal eyes
* Ametropia between -10D and +10D.

Exclusion Criteria:

* One pathological eye
* Prior ocular surgery
* Amblyopia, refraction larger than ±10D
* Corneal or retinal pathologies
* Systemic diseases (e.g. diabetes, multiple sclerosis, …)
* More than 5 months pregnant at the moment of testing
* Recent wear of hard contact lenses
* Epilepsy (if C-Quant is used).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal subjects
Sampling Method: Probability Sample
Enrollment: 1646 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
to obtain a predetermined number of valid ocular biometry measurements per participating site | 19 months
  The test that will be performed are the eye dominance, uncorrected and corrected distance visual acuity (UDVA and CDVA), (accommodation, ocular refraction (automatic refraction), spectacle refraction, axial length (optical, ultrasound), anterior segment biometry (anterior chamber depth), corneal topography (keratometry), contrast sensitivity (Pelli-Robson/ Sine Wave Contrast Test (SWCT), pupil size (gauge)), intraocular pressure, the VFQ-25 questionnaire and some demographic data (age, gender, ethnicity, eye color, highest education).
To obtain a predetermined number of valid visual function measurements per participating site | 19 months
  The tests that will be performed are the eye dominance, accommodation, uncorrected and spectacle corrected visual acuity (UCVA and SCVA), ocular refraction (automatic refraction), spectacle refraction, axial length (optical, ultrasound), anterior segment biometry (anterior chamber depth), corneal topography (keratometry), contrast sensitivity (Pelli-Robson/ Sine Wave Contrast Test (SWCT)), intraocular pressure, the VFQ-25 questionnaire and some demographic data (age, gender, ethnicity, eye color, highest education).

SECONDARY OUTCOMES:
Provide a reference database for research purposes | 19 Months
  Protocol foresees in inclusion optional tests:straylight measurement (using Oculus C-Quant,pupillometry,distance-corrected intermediate and near visual acuity(DCIVA and DCNVA,crystalline lens thickness,aberrometry,ORA measurements (IOPcc,IOPG,CRF,CH parameters.These tests may be added by the individual sites depending of the availability of equipment.A number of secondary parameters can also be derived from primary parameters using calculations (e.g.crystalline lens power, estimated aniseikonia,etc) or by analysis of the raw data of computer based tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jos Rozema, MSc PhD, Study Chair — Dept of Ophthalmology, Antwerp University Hospital. Edegem, Belgium; Marie-José Tassignon, MD PhD, Principal Investigator — Dept of Ophthalmology, Antwerp University Hospital. Edegem, Belgium; Sotiris Plainis, MSc PhD, Principal Investigator — Institute of Vision and Optics (IVO), University of Crete, School of Health Sciences, Heraklion Crete, Greece 71003
Locations (1):
- VISSUM - Instituto Oftalmológico de Alicante, Alicante, Spain, Spain

REFERENCES:
- [Derived] Zocher MT, Rozema JJ, Oertel N, Dawczynski J, Wiedemann P, Rauscher FG; EVICR.net. Biometry and visual function of a healthy cohort in Leipzig, Germany. BMC Ophthalmol. 2016 Jun 7;16:79. doi: 10.1186/s12886-016-0232-2. PMID 27268271